CLINICAL TRIAL: NCT06238869
Title: Multi-faceted Online Interventions to Promoting Mental Health in Children and Adolescents:a Population-based, Cluster-randomized Controlled Trial
Brief Title: Online Mental Health Interventions for Children and Adolescents (OMHICA)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Jiangsu Province Nanjing Brain Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 81725005-9
Record Dates: First submitted 2024-01-25; First posted 2024-02-02 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-01

CONDITIONS: Depression; Anxiety; Stress; Insomnia
Keywords: Computerized Cognitive Behavioral Therapy; Music Therapy; Health education; Acoustic features
MeSH Terms: conditions — Depression; Anxiety Disorders; Sleep Initiation and Maintenance Disorders; Health Education | interventions — Music Therapy

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Computerized Cognitive Behavioral Therapy (CCBT) (Experimental): The experimental group received a 4-week CCBT intervention, which consisted of completing 3 modules every week, each taking roughly 20 minutes.
  Interventions: Behavioral: Computerized Cognitive Behavioral Therapy
- Music Therapy(MT) (Experimental): All the participants of Music Therapy will be treated with 12 sessions (3 sessions per week),15 minutes each time, and conducted for 4 weeks.
  Interventions: Behavioral: Music Therapy
- Health education (Experimental): The health education group will conduct a series of mental health lectures through the WeChat Mini Program on a weekly basis, with each session lasting for 30 minutes, spanning over a duration of four weeks.
  Interventions: Behavioral: Health education
- Blank Control Group (No Intervention): All the participants in this group receive no intervention and undergo only psychological health screenings at designated time points.

INTERVENTIONS:
Behavioral: Computerized Cognitive Behavioral Therapy — CCBT (Computerized Cognitive Behavioral Therapy) is a unique approach to improving mental well-being. It utilizes computer-based cognitive and behavioral techniques to induce relaxation and regulate emotional responses by targeting specific brain regions. CCBT offers interactive and personalized interventions, empowering individuals to address mental health challenges like depression and anxiety. Its convenience and accessibility through digital platforms make it a practical choice for enhancing emotional well-being.
  Arms: Computerized Cognitive Behavioral Therapy (CCBT)
Behavioral: Music Therapy — Music Therapy can make peoples gradually relax via relaxing and soothing music, and regulate individual psychological emotions through the influence of music on individuals' cerebral cortex, hypothalamus and limbic system, further improve the mood of daily tension and anxiety.
  Arms: Music Therapy(MT)
Behavioral: Health education — Health education focuses on providing insights into adolescent mental health, offering practical coping strategies and behavior patterns. It emphasizes the crucial link between parental guidance and the well-being of adolescents. By fostering healthier psychological interactions, it cultivates an environment supportive of adolescent mental health, strengthens family support, and promotes comprehensive development in physical, mental, and cognitive aspects.
  Arms: Health education

SUMMARY:
Mental health has become an increasing concern, especially among children and adolescents in schools. However, not all individuals in mental suboptimal states require pharmacological treatment. With the development of internet technology, internet-based psychological therapy methods are considered to have tremendous potential and are being given significant attention. Simultaneously, due to their convenience, these approaches are widely applied. Computerized Cognitive Behavioral Therapy (CCBT) can achieve its therapeutic effect by improving activation patterns of the brain's internal networks to promote self-regulation. Music Therapy (MT) can make peoples gradually relax via relaxing and soothing music, and regulate individual psychological emotions through the influence of music on individuals' cerebral cortex, hypothalamus and limbic system, further improve the mood of daily tension and anxiety. Health Education works to provide parents with knowledge and information about mental health, aiming to help them better understand and support their own and their children's mental health, thereby improving parent-child relationships.

The study was designed as a randomized clinical trial with four groups, the CCBT group, the MT group, the Health Education group and the control group in children and adolescent .The CCBT group, the MT group, and the Health Education group all completed their interventions through online self-help therapy. The control group did not receive any intervention. Data collection was conducted by trained, certified and qualified personnel.

The mental health intervention is a crucial component of the "School-based Evaluation Advancing Response for Child Health (SEARCH)" cohort study, focusing on observing changes in the population undergoing the intervention within the cohort study.

DETAILED DESCRIPTION:
The online intervention study was a population-based, cluster-randomized controlled trial that aimed to evaluate the efficacy of various interventions promoting mental health in children and adolescent.

The CCBT intervention consisted of two components: (a) The participants were presented with 12 modules. All modules were based on the cognitive- behavioral model by Beck and informed by the updated procedures by J. Beck and Wright. Modules 1-2 introduce the definitions, symptoms, causes and basic cognitive models of depression and anxiety. Modules 3-6 describe how to identify cognitive distortions and deal with negative automatic thoughts in daily life. Modules 7-8 mainly focus on behavioral activation and dealing with intermediate beliefs. Modules 9-11 center on learning about structured problem-solving approaches and core beliefs. Module 12 describes a summary of treatment and relapse prevention. (b) After each module is completed, we send a notification of homework to the subjects, and their compliance is assessed by registering completed modules and homework. The experimental group received a 4-week CCBT intervention, which consisted of completing 3 modules every week, each taking roughly 20 minutes.

All the participants of Music Therapy will be treated with 12 sessions (3 sessions per week),15 minutes each time, and conducted for 4 weeks. The MT is mainly divided into three stages, and each stage has a topic. The topic of each stage as follow: physical and mental relaxation stage: learning the whole body and mind relaxation mode from breathing to muscle; nature imagination stage: guiding music imagination; internal self-exploration: excavating the positive experience and positive potential of the listener and adopting resource orientation for psychological intervention.

The health education group will conduct a series of mental health lectures through the WeChat Mini Program on a weekly basis, with each session lasting for 30 minutes, spanning over a duration of four weeks. The themes of mental health lectures were:1.Parents communicate well with their children, and they thrive in the sun;2.Three effective increments in the growth of adolescents;3.early identification and intervention of adolescent emotional disorders;4.brain and emotions. While the control group did not receive any intervention during the same time.

ELIGIBILITY:
Inclusion Criteria:

* Willing elementary students, with parental consent, to undergo mental health screenings and engage in subsequent mental health activities.
* Ages between 11 and 19.
* Participants who can operate a mobile phone and can read and receive messages on "WeChat".

Exclusion Criteria:

* Participants with self-reported lifetime suicide attempts, active self-harm, or active suicidal ideation with intent will be excluded from the study.
* Have a diagnosis by a clinician of bipolar disorder, substance use disorder, or any psychotic disorder including schizophrenia
* Individuals who are incapable of understanding or completing study procedures and digital intervention, as determined by the participant, patient/legal guardian, healthcare provider, or clinical research team, will be excluded.

Ages: 11 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 7000 (Estimated)
Dates: Start 2024-01-26 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in DASS-depression detection rate | Baseline, week 4 and week 28
  Change from baseline in the screening rate of depressive symptoms assessed by The Depression Anxiety Stress Scale within the population.
Change from baseline in DASS-anxiety detection rate | Baseline, week 4 and week 28
  Change from baseline in the screening rate of anxiety symptoms assessed by The Depression Anxiety Stress Scale within the population.
Change from baseline in DASS-stress detection rate | Baseline, week 4 and week 28
  Change from baseline in the screening rate of stress symptoms assessed by The Depression Anxiety Stress Scale within the population.
Change from baseline in Insomnia Severity Index (ISI) questionnaire insomnia detection rate | Baseline, week 4 and week 28
  Insomnia Severity Index (ISI) questionnaire insomnia detection rate refers to the rate at which insomnia is identified or detected based on responses from the ISI questionnaire. The ISI is a validated tool used to assess insomnia symptom severity and their impact on daily functioning. The detection rate indicates the proportion of individuals in a population or sample whose ISI questionnaire responses indicate the presence of insomnia.

SECONDARY OUTCOMES:
Change from baseline in depressive symptom assessed by The Depression Anxiety Stress Scale (DASS) at week 4, week 8, and week 28. | Baseline, week 4 and week 28
  The DASS Depression scale, with scores ranging from 0 to 42, is interpreted as follows for different severity levels of depression: normal (0-9), mild (10-13), moderate (14-20), severe (21-27), and extremely severe (28+).
Change from baseline in anxiety symptom assessed by The Depression, Anxiety and Stress Scale (DASS)at week 4, week 8, and week 28. Stress Scale (DASS) at week 4, week 8, and week 28. | Baseline, week 4 and week 28
  The DASS Anxiety scale, also with scores ranging from 0 to 42, has the following grading criteria: normal (0-7), mild (8-9), moderate (10-14), severe (15-19), and extremely severe (20+).
Change from baseline in stress symptom assessed by The Depression Anxiety Stress Scale (DASS) at week 4, week 8, and week 28. | Baseline, week 4 and week 28
  The DASS Stress scale, which also has scores ranging from 0 to 42, the grading criteria are as follows: normal (0-14), mild (15-18), moderate (19-25), severe (26-33), and extremely severe (34+).
Change from baseline in insomnia symptoms assessed by the Insomnia Severity Index (ISI; range: 0-28) at week 4, week 8, and week 28. | Baseline, week 4 and week 28
  The total scores of these questionnaires were interpreted as follows: normal (0-7), mild (8-14), moderate (15-21), and severe (22-28) insomnia.
Change from baseline in acoustic features. | Baseline, week 4 and week 28
  Participants will record videos prior to beginning intervention (baseline) and after completing intervention (week 4, week 8, and week 28). Participants read the poem "The North Wind and the Sun" in a quiet environment and recorded it to obtain the voice snippets. Acoustic features are a set of indicators that can reflect an individual's emotional state. The indicators include LOGenergy, zero-crossing rate, fband, spectralRollOff, melspec spectral flux, centroid, maxPos, minPos mfcc, voiceProb F0, F0env etc.
Change from baseline in the facial expression features measured. | Baseline and week 28
  Participants will record audio prior to beginning intervention (baseline) and after completing intervention (week 4, week 8 and week 28). Participants were given a series of dynamic facial expressions by answering short on-screen questions and tapping a record video button on the screen. Facial features are a set of indicators that can reflect an individual's emotional state, including eye characteristics, facial action unit, head features, deformation shape parameter. Previous studies have found that the more severe the depressive symptoms, the sadder the expression and the less the patient smiles. As depressed mood improves, depressed expressions and the patient's range of body movements can improve accordingly.
Change from baseline in the Strengths and Difficulties Situation assessed by Strengths and Difficulties Questionnaire (SDQ). | Baseline and week 28
  SDQ includes five scales of five items each: emotional symptoms, conduct problems, hyperactivity, peer problems, and prosocial behavior. Each subscale comprises 5 questions with response options of 0,1, and 2 points. The score range for each subscale is from 0 to 10 points. A higher score on each subscale indicates more severe issues in that particular aspect.
Change from baseline in resting-state magnetic resonance imaging (MRI), diffusion tensor imaging (DTI) and structural (T1-weighted) imaging at baseline and week 4 | Baseline and week 4
  Participants will undergo MRI scans before (week 0) and after completing (week 4) the treatment. This allows for a comprehensive examination of changes in functional activity, DTI and structural changes in the brain between baseline and weeks 4.
Change in the influence of the family environment on the individual, as assessed by the Family Environment Scale (FES), from baseline to week 4 and week 28. | Baseline and week 28
  The FES scale has seven factors, which are intimacy, conflict, success, culture, entertainment, organization, control, and these 7 dimensions measure the influence of family on individuals.
The change from baseline in internet addiction symptom was assessed by the Internet Addiction Scale at week 4 and week 28. | Baseline and week 28
  The Internet Addiction Scale has five factors, namely compulsive Internet use, Internet addiction withdrawal reaction, Internet addiction tolerance, time management problems, interpersonal and health problems. The higher the total score, the deeper the degree of Internet addiction.
The change from baseline in the implementation of NSSI behaviors was assessed by Ottawa Self-injury Inventory (OSI) at week 4 and week 28. | Baseline and week 28
  OSI is used to assess the prevalence of NSSI, including the frequency, concealment and reasons for NSSI.
The change from baseline in the victimization of bullying since enrollment was assessed by Delaware Bullying Victimization Scale (DBVS) at week 4 and week 28. | Baseline and week 28
  DBVS was used to assess the bullying behaviors, including physical bullying, relational bullying, verbal bullying and cyberbullying. The total scale score is the sum of the item scores, with higher total scores indicating more severe bullying.
The change from baseline in childhood traumatic experiences was assessed by Childhood Trauma Questionnaire-28 item Short Form(CTQ-SF) at week 4 and week 28. | Baseline and week 28
  CTQ-SF contained four factors: emotional abuse, physical abuse, emotional neglect and physical neglect. Emotional neglect ≥15, physical neglect ≥10, emotional abuse ≥13, and physical abuse ≥10.
The change from baseline in food addiction symptom was assessed by Modified Yale Food Addiction Scale (mYFAS) at week 4 and week 28. | Baseline and week 28
  The mYFAS is used to assess food addiction symptoms for diet-related impairment and distress. The scale is assessed on an 8-point scale ranging from 0 (never) to 7 (daily).

CONTACTS AND LOCATIONS:
Overall Officials: Fei Wang, Ph.D, Study Chair — Nanjing Brain Hospital, Nanjing Medical University
Locations (1):
- Affiliated Brain Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No